CLINICAL TRIAL: NCT03797989
Title: VAC069: A Clinical Study to Assess the Safety and Feasibility of Controlled Blood-stage Plasmodium Vivax Human Malaria Infection Through Experimental Inoculation of Cryopreserved Infected Erythrocytes in Healthy Malaria-naïve UK Adults
Brief Title: VAC069: A Study of Blood-stage Controlled Human P. Vivax Infection
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: VAC069
Record Dates: First submitted 2018-11-29; First posted 2019-01-09 (Actual); Results first posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2023-03

CONDITIONS: Malaria, Vivax
MeSH Terms: conditions — Malaria, Vivax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Phase A: Group 1 (Experimental): Each volunteer will receive one vial of P. vivax infected inoculum (parasitised red blood cells) at the first blood-stage controlled human malaria infection (CHMI). The optimal dose will be determined following the first CHMI and the selected dose will be administered to all volunteers (Groups 1-3) at both the second and third CHMI.
  Interventions: Biological: P. vivax infected inoculum (parasitised red blood cells)
- Phase A: Group 2 (Experimental): Each volunteer will receive a fifth of a vial (1:5 dilution) of P. vivax infected inoculum (parasitised red blood cells) at the first blood-stage controlled human malaria infection (CHMI). The optimal dose will be determined following the first CHMI and the selected dose will be administered to all volunteers (Groups 1-3) at both the second and third CHMI.
  Interventions: Biological: P. vivax infected inoculum (parasitised red blood cells)
- Phase A: Group 3 (Experimental): Each volunteer will receive one twentieth of a vial (1:20 dilution) of P. vivax infected inoculum (parasitised red blood cells) at the first blood-stage controlled human malaria infection (CHMI). The optimal dose will be determined following the first CHMI and the selected dose will be administered to all volunteers (Groups 1-3) at both the second and third CHMI.
  Interventions: Biological: P. vivax infected inoculum (parasitised red blood cells)
- Phase B: Group 4 (Experimental): The six volunteers from Groups 1, 2 and 3 in will undergo secondary challenge using the optimal inoculum, as determined in Phase A of the study. They will constitute 'Group 4' in Phase B. This will occur approximately eight months (and up to nine months) later after their primary challenge.
  Interventions: Biological: P. vivax infected inoculum (parasitised red blood cells)
- Phase B: Group 6 (Experimental): Three new malaria naïve volunteers will be recruited to undergo primary challenge using the optimal inoculum, as determined in Phase A of the study. They will act as controls to Group 4.
  Interventions: Biological: P. vivax infected inoculum (parasitised red blood cells)
- Phase C: Group 5 (Experimental): The six volunteers from Group 4 in Phase B will undergo tertiary challenge, again using the optimal inoculum as determined in Phase A, and will constitute Group 5 in Phase C. This will occur approximately sixteen months (and up to twenty months) later after their secondary challenge.
  Interventions: Biological: P. vivax infected inoculum (parasitised red blood cells)
- Phase C: Group 7 (Experimental): The three volunteers from Group 6 who underwent primary challenge in Phase B undergo secondary challenge, again using the optimal inoculum as determined in Phase A, and will now form Group 7 in Phase C. This will occur approximately six months (and up to nine months) later after their primary challenge.
  Interventions: Biological: P. vivax infected inoculum (parasitised red blood cells)
- Phase C: Group 9 (Experimental): Four to eight new malaria-naïve volunteers will be recruited to undergo primary challenge using the optimal inoculum, as determined in Phase A of the study. They will act as controls for Groups 5 and 7.
  Interventions: Biological: P. vivax infected inoculum (parasitised red blood cells)
- Phase D: Group 8 (Experimental): The three volunteers from Group 7 in Phase C will undergo tertiary challenge, again using the optimal inoculum as determined in Phase A, and will constitute Group 8 in Phase D. This will occur approximately five months (and up to ten months) after their secondary challenge.
  Interventions: Biological: P. vivax infected inoculum (parasitised red blood cells)
- Phase D: Group 10 (Experimental): The four to eight volunteers from Group 9 in Phase C will undergo secondary challenge, using the optimal inoculum as determined in Phase A, and form Group 10 in Phase D. This will occur approximately six months (and up to nine months) later after their primary challenge.
  Interventions: Biological: P. vivax infected inoculum (parasitised red blood cells)
- Phase D: Group 12 (Experimental): Four to eight new malaria-naïve volunteers will be recruited to undergo primary challenge using the optimal inoculum, as determined in Phase A of the study. They will act as controls for Groups 8 and 10.
  Interventions: Biological: P. vivax infected inoculum (parasitised red blood cells)
- Phase E: Group 13 (Experimental): Volunteers from Groups 10 and 12 who completed at least one P. vivax CHMI in Phase D will be re-enrolled into Group 13 to undergo repeat heterlogous CHMI with P. falciparum in Phase E. This will occur occur approximately 12 months after their last P. vivax challenge.
  Interventions: Biological: P. vivax infected inoculum (parasitised red blood cells)

INTERVENTIONS:
Biological: P. vivax infected inoculum (parasitised red blood cells) — In the first controlled human malaria infection (CHMI, Phase A), inoculation of parasitised red blood cells will be at three different doses (1 vial, 1:5 dilution, 1:20 dilution). The optimal inoculation dose will then be selected and administered to all participants in each of the second and third CHMI.

SUMMARY:
This is a clinical study to assess the safety and feasibility of Plasmodium vivax (P. vivax) controlled blood-stage human malaria infection (CHMI), by inoculation using a newly created source of P. vivax malaria-infected blood.

25 healthy malaria-naïve UK volunteers, aged 18 - 50, will be recruited through the five phases of the study at the CCVTM, Oxford. Volunteers will undergo primary, secondary and tertiary P. vivax blood-stage challenges, which will be induced by injection of P. vivax infected blood. After the first challenge, the optimal dose for blood-stage CHMI will be selected and used for the second and third challenges. Through each challenge period, volunteers will have blood taken at regular intervals to measure the parasite growth, quantify the sexual parasite forms and assess the immune response to P. vivax infection. Transmission of P. vivax from volunteers to the Anopheline mosquito vectors will also be assessed.

In each challenge, following diagnosis, volunteers will be treated with a standard antimalarial course of oral artemether-lumefantrine (Riamet), given over 60 hours. Volunteers who take part in this study will be involved in the trial for approximately 2 years, receiving each of the three challenges at intervals of approximately 5 (and up to 9) months. Volunteers will be followed for 3 months after their last challenge.

DETAILED DESCRIPTION:
This study aims primarily to assess the safety and feasibility of controlled blood-stage human P. vivax malaria infection. This will be the first time that this source of P. vivax infected blood will be utilised and the first P. vivax bloodstage CHMI in Europe. If demonstrated to be safe, it is intended that this parasitised blood bank be used in future CHMI studies to evaluate candidate vaccines.

This study will also assess parasite growth, including quantifying the sexual-stage parasites in the blood, as well as the transmission of P. vivax from volunteers to the Anopheline mosquito vectors and the immune responses in primary, secondary and tertiary P. vivax blood-stage challenge, as further secondary aims. Natural immunity to P. vivax is acquired over time, following repeated exposure. Repeated blood-stage challenge would improve understanding of how the human immune response to P. vivax infected is acquired, and how parasite growth changes in a second or third exposure. Repeated challenges can also be used to test if potential vaccine candidates can protect against repeated malaria infection. If proven to be safe and feasible in this study, this will provide a basis for conducting P. vivax blood-stage re-challenge studies for evaluation of new vaccine candidates.

The study is funded through The Wellcome Trust and MultiViVax, a European Commission Horizon 2020 funded project.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult aged 18 to 50 years.
* Red blood cells positive for the Duffy antigen/chemokine receptor (DARC).
* Normal serum levels of Glucose-6-phosphate dehydrogenase (G6PDH).
* Negative haemoglobinopathy screen
* Able and willing (in the Investigator's opinion) to comply with all study requirements.
* Willing to allow the Investigators to discuss the volunteer's medical history with their General Practitioner.
* Women only: Must practice continuous effective contraception for the duration of the clinic visits (first 3 months post-CHMI).
* Agreement to permanently refrain from blood donation
* Written informed consent to participate in the trial.
* Reachable (24/7) by mobile phone during the period between CHMI and completion of all antimalarial treatment.
* Willing to take a curative anti-malarial regimen following CHMI.
* Willing to reside in Oxford for the duration of the study, until antimalarials have been completed.
* Answer all questions on the informed consent quiz correctly.

Exclusion Criteria:

* History of clinical malaria (any species).
* Travel to a clearly malaria endemic locality during the study period or within the preceding six months.
* Use of systemic antibiotics with known antimalarial activity within 30 days of CHMI (e.g.trimethoprim-sulfamethoxazole, doxycycline, tetracycline, clindamycin, erythromycin, fluoroquinolones and azithromycin).
* Haemoglobin <120 g/L for a female volunteer or <130 g/L for a male volunteer prior to primary CHMI. (However, for enrolment into secondary and tertiary CHMIs slightly lower haemoglobin values (≤0.5 g/L) will be permitted at the discretion of the Investigator, to account for the blood volume donated during the previous CHMI).
* Receipt of immunoglobulins within the three months prior to enrolment.
* Receipt of blood transfusion at any time in the past.
* Peripheral venous access unlikely to allow twice daily blood testing (as determined by the Investigator).
* Receipt of an investigational product in the 30 days preceding enrolment, or planned receipt during the study period.
* Prior receipt of an investigational vaccine likely to impact on interpretation of the trial data or the P. vivax parasite as assessed by the Investigator.
* Planned receipt of a COVID-19 vaccine between 2 weeks before the day of CHMI until completion of antimalarial treatment
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed).
* History of allergic disease or reactions likely to be exacerbated by malaria infection.
* Pregnancy, lactation or intention to become pregnant during the study.
* Use of medications known to cause prolongation of the QT interval and existing contraindication to the use of Malarone.
* Use of medications known to have a potentially clinically significant interaction with Riamet and Malarone.
* Any clinical condition known to prolong the QT interval.
* History of cardiac arrhythmia, including clinically relevant bradycardia.
* Disturbances of electrolyte balance, e.g. hypokalaemia or hypomagnesaemia.
* Family history of congenital QT prolongation or sudden death.
* Contraindications to the use of both of the proposed anti-malarial medications Riamet and Malarone.
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
* History of serious psychiatric condition that may affect participation in the study.
* Any other serious chronic illness requiring hospital specialist supervision.
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 25 standard UK units every week.
* Suspected or known injecting drug abuse in the 5 years preceding enrolment.
* Hepatitis B surface antigen (HBsAg) detected in serum.
* Seropositive for hepatitis C virus (antibodies to HCV) at screening or at C-7 (unless has taken part in a prior hepatitis C vaccine study with confirmed negative HCV antibodies prior to participation in that study, and negative HCV RNA PCR at screening for this study).
* Positive family history in both 1st AND 2nd degree relatives < 50 years old for cardiac disease.
* Volunteers unable to be closely followed for social, geographic or psychological reasons.
* Any clinically significant abnormal finding on biochemistry or haematology blood tests, urinalysis or clinical examination. In the event of abnormal test results, confirmatory repeat tests will be requested.
* Any other significant disease, disorder, or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.
* Inability of the study team to contact the volunteer's GP to confirm medical history and safety to participate.
* Additional exclusion criteria for Groups 6-13: Body weight <50Kg, as measured at screening

Exclusion criteria on day of CHMI:

* Acute disease, defined as moderate or severe illness with or without fever.
* Current COVID-19 infection, defined as ongoing symptoms with positive COVID-19 PCR swab test taken during current illness or positive COVID-19 PCR swab test within preceding 14 days without symptoms.
* Pregnancy.
* Potential volunteers who are due to have a COVID-19 vaccine in the period between 2 weeks before the day of malaria challenge and expected time of completion of malaria treatment will not be enrolled (estimate up to 3 weeks after day of challenge based on experience in this study to date). If a volunteer receives an appointment for COVID-19 vaccination after they have undergone malaria challenge but before reaching malaria diagnosis criteria, they will be advised to delay their COVID-19 vaccination until after reaching malaria diagnostic criteria and completion of antimalarial treatment. If a participant does not wish to delay their COVID-19 vaccination, they will be treated with antimalarial treatment at that time point and withdrawn from the study but will be encouraged to complete follow-up for safety.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela M Minassian, MBBS MA DPhil MRCP FRCPath, Principal Investigator — University of Oxford
Locations (1):
- Centre for Clinical Vaccinology & Tropical Medicine, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Derived] Hou MM, Harding AC, Barber NM, Kundu P, Bach FA, Salkeld J, Themistocleous Y, Greenwood NM, Cho JS, Barrett JR, Nugent FL, Rawlinson TA, Hodgson SH, Khozoee B, Mac Lochlainn DJ, Cowan RE, Poulton ID, Baker M, Kingham L, Mitton CH, Platt A, Lopez Ramon R, Ramos Lopez F, Thomas M, Skinner K, Quinkert D, Pipini D, Lias AM, Bardelli M, Edwards NJ, Donnellan FR, Biswas S, Rayner JC, Nielsen CM, Silk SE, Draper SJ, Nahrendorf W, Spence PJ, Minassian AM. Development of clinical immunity to Plasmodium vivax following repeat controlled human malaria infection. Nat Commun. 2025 Sep 25;16(1):8385. doi: 10.1038/s41467-025-63104-y. PMID 40998768
- [Derived] Bach FA, Munoz Sandoval D, Mazurczyk M, Themistocleous Y, Rawlinson TA, Harding AC, Kemp A, Silk SE, Barrett JR, Edwards NJ, Ivens A, Rayner JC, Minassian AM, Napolitani G, Draper SJ, Spence PJ. A systematic analysis of the human immune response to Plasmodium vivax. J Clin Invest. 2023 Oct 16;133(20):e152463. doi: 10.1172/JCI152463. PMID 37616070
- [Derived] Hou MM, Barrett JR, Themistocleous Y, Rawlinson TA, Diouf A, Martinez FJ, Nielsen CM, Lias AM, King LDW, Edwards NJ, Greenwood NM, Kingham L, Poulton ID, Khozoee B, Goh C, Mac Lochlainn DJ, Salkeld J, Guilotte-Blisnick M, Huon C, Mohring F, Reimer JM, Chauhan VS, Mukherjee P, Biswas S, Taylor IJ, Lawrie AM, Cho JS, Nugent FL, Long CA, Moon RW, Miura K, Silk SE, Chitnis CE, Minassian AM, Draper SJ. Impact of a blood-stage vaccine on Plasmodium vivax malaria. medRxiv [Preprint]. 2022 May 30:2022.05.27.22275375. doi: 10.1101/2022.05.27.22275375. PMID 35664997
- [Derived] Minassian AM, Themistocleous Y, Silk SE, Barrett JR, Kemp A, Quinkert D, Nielsen CM, Edwards NJ, Rawlinson TA, Ramos Lopez F, Roobsoong W, Ellis KJ, Cho JS, Aunin E, Otto TD, Reid AJ, Bach FA, Labbe GM, Poulton ID, Marini A, Zaric M, Mulatier M, Lopez Ramon R, Baker M, Mitton CH, Sousa JC, Rachaphaew N, Kumpitak C, Maneechai N, Suansomjit C, Piteekan T, Hou MM, Khozoee B, McHugh K, Roberts DJ, Lawrie AM, Blagborough AM, Nugent FL, Taylor IJ, Johnson KJ, Spence PJ, Sattabongkot J, Biswas S, Rayner JC, Draper SJ. Controlled human malaria infection with a clone of Plasmodium vivax with high-quality genome assembly. JCI Insight. 2021 Dec 8;6(23):e152465. doi: 10.1172/jci.insight.152465. PMID 34609964

RESULTS

PARTICIPANT FLOW:
Period: VAC069A
Arm/Group | Phase A: Group 1 | Phase A: Group 2 | Phase A: Group 3 | Phase B: Group 4 | Phase B: Group 6 | Phase C: Group 5 | Phase C: Group 7 | Phase C: Group 9 | Phase D: Group 8 | Phase D: Group 10 | Phase D: Group 12 | Phase E: Group 13
Started | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: VAC069B
Arm/Group | Phase A: Group 1 | Phase A: Group 2 | Phase A: Group 3 | Phase B: Group 4 | Phase B: Group 6 | Phase C: Group 5 | Phase C: Group 7 | Phase C: Group 9 | Phase D: Group 8 | Phase D: Group 10 | Phase D: Group 12 | Phase E: Group 13
Started | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: VAC069C
Arm/Group | Phase A: Group 1 | Phase A: Group 2 | Phase A: Group 3 | Phase B: Group 4 | Phase B: Group 6 | Phase C: Group 5 | Phase C: Group 7 | Phase C: Group 9 | Phase D: Group 8 | Phase D: Group 10 | Phase D: Group 12 | Phase E: Group 13
Started | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 7 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 7 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: VAC069D
Arm/Group | Phase A: Group 1 | Phase A: Group 2 | Phase A: Group 3 | Phase B: Group 4 | Phase B: Group 6 | Phase C: Group 5 | Phase C: Group 7 | Phase C: Group 9 | Phase D: Group 8 | Phase D: Group 10 | Phase D: Group 12 | Phase E: Group 13
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 7 | 4 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 7 | 4 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: VAC069E
Arm/Group | Phase A: Group 1 | Phase A: Group 2 | Phase A: Group 3 | Phase B: Group 4 | Phase B: Group 6 | Phase C: Group 5 | Phase C: Group 7 | Phase C: Group 9 | Phase D: Group 8 | Phase D: Group 10 | Phase D: Group 12 | Phase E: Group 13
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only study groups with new participants are included in this baseline analysis population. Groups 4, 5, 7, 8 and 10 consist of volunteers who were previously enrolled in a preceding group in this study and have completed one or two previous phases in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase A: Group 1 | Phase A: Group 2 | Phase A: Group 3 | Phase B: Group 6 | Phase C: Group 9 | Phase D: Group 12 | Total
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 7 | 4 | 19
Age, Continuous [Median (Full Range); unit: years] | 32 [31 to 33] | 25.5 [25 to 26] | 22.5 [18 to 27] | 26 [23 to 29] | 27 [22 to 48] | 25.5 [21 to 28] | 26 [18 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 1 | 4 | 2 | 9
  Male | 1 | 1 | 2 | 1 | 3 | 2 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2 | 1 | 1 | 2 | 4 | 4 | 14
  Arab | 0 | 1 | 0 | 0 | 1 | 0 | 2
  Asian | 0 | 0 | 1 | 0 | 1 | 0 | 2
  Mixed - White and Asian | 0 | 0 | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United Kingdom | 2 | 2 | 2 | 2 | 7 | 4 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events
Time Frame: 36 months
Population: Number of SAEs occuring during study period
Measure: Count of Participants; unit: Participants
Groups:
- Primary P. Vivax CHMI: Malaria naive volunteers who underwent primary controlled human malaria infection (CHMI) with blood-stage P. vivax during phases VAC069A to VAC069D of the study.
Arm/Group | Primary P. Vivax CHMI
Number analyzed (Participants) | 19
Participants | 1

2. Primary Outcome: Number of Participants Who Developed Infection/Reached Diagnosis Criteria, Used to Select the Optimal Inoculation Dose to Take Forward to Future P. Vivax CHMI Studies Based on a Protocol-specified Algorithm
Description: Choosing the optimal inoculation dose to take forward to future P. vivax CHMI studies will be decided based on the following algorithm:
  Ideal choice = the first group (2/2 volunteers) to reach diagnosis criteria (within 21 days). N.B. If both volunteers in Group 1 develop infection AND both volunteers in Group 2 (or 3) reliably develop infection within 5 days of Group 1 (and within the 21-day window) then the lowest dose group should be chosen.
Time Frame: 3 months
Population: All 6 volunteers who underwent primary CHMI during phase VAC069A of the study developed malaria infection and reached diagnostic criteria. An inoculation dose of 1:10 dilution of 1 vial of inoculum per volunteer was chosen for subsequent phases of the study VAC069B to VAC069D.
Measure: Number; unit: Participants who developed infection
Arm/Group | Phase A: Group 1 | Phase A: Group 2 | Phase A: Group 3
Number analyzed (Participants) | 2 | 2 | 2
Participants who developed infection | 2 | 2 | 2

3. Primary Outcome: Feasibility of Primary P. Vivax Blood-stage CHMI as Measured by Successful Infection (Development of Detectable Persistent Parasitaemia by Thick Film and qPCR +/- Clinical Symptoms)
Description: Number of participants developing detectablable parasitaemia during primary CHMI with P. vivax (PvW1 clone)
Time Frame: 36 months
Population: All volunteers undergoing primary controlled human malaria infection with P. vivax (PvW1 clone)
Measure: Count of Participants; unit: Participants
Arm/Group | Primary P. Vivax CHMI
Number analyzed (Participants) | 19
Participants | 19

4. Secondary Outcome: Safety of Secondary and Tertiary P. Vivax Controlled Blood-stage CHMI as Measured by (S)AE Occurrences
Time Frame: 36 months
Population: Number of SAEs occuring during study period
Measure: Count of Participants; unit: Participants
Groups:
- Secondary P. Vivax CHMI: Volunteers who completed one P. vivax CHMI in the preceding phase of the study, underwent secondary CHMI with P. vivax during phases VAC069B to VAC069D of the study.
- Tertiary P. Vivax CHMI: Volunteers who completed their second P. vivax CHMI in the preceding phase of the study, underwent tertiary CHMI with P. vivax during phases VAC069C and VAC069D of the study.
- VAC069E - P. Falciparum CHMI: Volunteers who completed primary or secondary P. vivax CHMI in phase VAC069D, underwent repeat heterlogous CHMI with P. falciparum in VAC069E.
Arm/Group | Secondary P. Vivax CHMI | Tertiary P. Vivax CHMI | VAC069E - P. Falciparum CHMI
Number analyzed (Participants) | 12 | 2 | 6
Participants | 0 | 0 | 0

5. Secondary Outcome: Immune Response to Primary, Secondary and Tertiary P. Vivax Pre-treatment
Description: As measured by antibody, B cell and T cell responses through experimental injection of P. vivax infected erythrocytes
Time Frame: 36 months
Reporting Status: Not Posted

6. Secondary Outcome: Gametocytaemia
Description: As measured by qPCR in primary, secondary and tertiary P. vivax blood-stage CHMI.
Time Frame: 36 months
Reporting Status: Not Posted

7. Secondary Outcome: Feasibility of Secondary and Tertiary P. Vivax Controlled Blood-stage CHMI as Measured by Successful Infection (Development of Detectable Persistent Parasitaemia by Thick Film and qPCR +/- Clinical Symptoms)
Time Frame: 36 months
Reporting Status: Not Posted

8. Secondary Outcome: Transmissibility of Gametocytes From the Infected Volunteer to Anopheline Mosquito Vector, Which Will be Assesed by Direct Membrane Feeding Assays (DMFA)
Time Frame: 36 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected from day of malaria challenge (CHMI) until 3 months after each challenge.
Arm/Group | Primary P. Vivax CHMI | Secondary P. Vivax CHMI | Tertiary P. Vivax CHMI | VAC069E - P. Falciparum CHMI
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/12 | 0/2 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/19 | 0/12 | 0/2 | 0/6
Other Adverse Events (participants affected / at risk) | 12/19 | 2/12 | 1/2 | 2/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Primary P. Vivax CHMI (N=19) | Secondary P. Vivax CHMI (N=12) | Tertiary P. Vivax CHMI (N=2) | VAC069E - P. Falciparum CHMI (N=6)
Upper limb fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 — Fracture of arm following road traffic accident
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Primary P. Vivax CHMI (N=19) | Secondary P. Vivax CHMI (N=12) | Tertiary P. Vivax CHMI (N=2) | VAC069E - P. Falciparum CHMI (N=6)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Tooth infection (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Stress (Psychiatric disorders) | 1 | 0 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/89/NCT03797989/Prot_SAP_000.pdf